CLINICAL TRIAL: NCT03326817
Title: A Soft Robotics Approach Towards Finger Joint Deformities in Rheumatic Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2017/00386
Record Dates: First submitted 2017-10-24; First posted 2017-10-31 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2017-09

CONDITIONS: Osteoarthritis
Keywords: Degenerative Arthritis, Rheumatic Diseases
MeSH Terms: conditions — Osteoarthritis; Rheumatic Diseases | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Comparing the control group and intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): This group will receive standard care.
  Interventions: Other: Control Group
- Soft Robotic Glove Group (Experimental): This group will receive standard care and soft robotic therapy (continuous passive motion device developed by National University of Singapore).
  Interventions: Device: Soft Robotic Glove Group

INTERVENTIONS:
Other: Control Group — Patients receive standard care
  Arms: Control Group
Device: Soft Robotic Glove Group — This group will receive standard care and soft robotic therapy (continuous passive motion device developed by National University of Singapore).
  Arms: Soft Robotic Glove Group

SUMMARY:
The study is to investigate the effect of a soft robotic glove approach providing continuous passive motion of fingers (flexion and extension) on degenerative arthritis patients. The approach may help reduce pain, maintain mobility and flexibility and to improve hand function.

DETAILED DESCRIPTION:
The aim is to investigate the effect of soft robotic gloves in providing continuous passive motion of the fingers (finger flexion and extension) of degenerative arthritis patients, for the purpose of providing pain relief and alleviating stiffness at the finger joints. Specifically, we intend to 1) observe the changes in range of motion of the fingers using the Total Active Motion (TAM) measure; 2) observe the changes in grip strength and pinch strength; and 3) record changes in the patients' perception of performance in activities of daily living using the Canadian Occupational Performance Measure (COPM).

The hypothesis is that a soft robotics approach in providing continuous passive motion of the finger joints of degenerative arthritis patients can reduce pain, maintain mobility and flexibility of the joints, and to improve hand function. The soft robotics approach and the standard hand therapy is better than the standard hand therapy alone.

The proposed soft robotic glove is capable of providing continuous passive motion (flexion and extension) of the fingers, and in addition, it is also designed to be portable and easy to operate, with minimal supervision. It is aimed at the home therapy of degenerative arthritis patients. In this study, by using the soft robotic glove and in observing changes in finger range of motion, grip and pinch strength, as well as perception of performance in daily activities. This is important in establishing this device as a viable means to ultimately slow down the progression of degenerative arthritis, and to significantly improve the patients' abilities in carrying out activities of daily living, which had been impaired by degenerative arthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 30-90 years regardless of race
2. Osteoarthritis of the hand (Consistent with ACR criteria 1990)
3. Ability to pay attention and maintain supported sitting for 45 mins continuously
4. Able to give own consent
5. Able to comprehend and follow commands (Abbreviated Mental Test >= 7)

Exclusion Criteria:

1. Inflammatory arthritis (e.g. rheumatoid arthritis), trigger fingers, carpal tunnel syndrome (by symptoms), finger contractures
2. Recent steroid injections in the wrist/hand joints within the past 3 months
3. Anti-inflammatory drugs (e.g. non-steroidal anti-inflammatory drugs or oral steroid) in the past 1 month
4. Old stroke and/or spasticity affecting the upper limbs
5. Epilepsy for the last 6 months as of the date of recruitment
6. Poor skin conditions which would hamper donning robotic gloves
7. Pregnancy

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-03-14 (Actual)

PRIMARY OUTCOMES:
Change in fingers' Total Active Motion | Week 1 baseline assessment and Week 11 post intervention assessment
  Measure hand range of motion in which the sum of the extension at the metacarpophalangeal (MCP), proximal interphalangeal (PIP), and distal interphalangeal (DIP) joints is subtracted from the total achievable flexion of the same joints. Unit: Degree
Change in grip and pinch strength | Week 1 baseline assessment and Week 11 post intervention assessment
  Measure hand strength. Unit: g/kg

SECONDARY OUTCOMES:
Change in patient's Canadian Occupational Performance Measure | Week 1 baseline assessment and Week 11 post intervention assessment.
  Identify issues of personal importance to the patient and to detect changes in a patient's self-perception of occupational performance over time.

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Salter RB, Hamilton HW, Wedge JH, Tile M, Torode IP, O'Driscoll SW, Murnaghan JJ, Saringer JH. Clinical application of basic research on continuous passive motion for disorders and injuries of synovial joints: a preliminary report of a feasibility study. J Orthop Res. 1984;1(3):325-42. doi: 10.1002/jor.1100010313. PMID 6481515
- [Result] Kitay GS, Koren MJ, Helfet DL, Parides MK, Markenson JA. Efficacy of combined local mechanical vibrations, continuous passive motion and thermotherapy in the management of osteoarthritis of the knee. Osteoarthritis Cartilage. 2009 Oct;17(10):1269-74. doi: 10.1016/j.joca.2009.04.015. Epub 2009 May 4. PMID 19433134
- [Result] Kjeken I, Dagfinrud H, Slatkowsky-Christensen B, Mowinckel P, Uhlig T, Kvien TK, Finset A. Activity limitations and participation restrictions in women with hand osteoarthritis: patients' descriptions and associations between dimensions of functioning. Ann Rheum Dis. 2005 Nov;64(11):1633-8. doi: 10.1136/ard.2004.034900. Epub 2005 Apr 13. PMID 15829571